CLINICAL TRIAL: NCT07054450
Title: Patient With Cervical Radiculopathy - Complete Assessment and Rehabilitation
Brief Title: Assessment and Rehabilitation in Cervical Radiculopathy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Filantropia Hospital (Other)
Responsible Party: Principal Investigator, Diana Kamal, PhD, Filantropia Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FilantropiaH
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Cervical Radicular Pain; Spondyloarthritis (SA); Neuropathic Pain Management; Quality of Life (QOL)
Keywords: cervical radiculopathy; physical medicine and rehabilitation; quality of life; nutraceutical treatment
MeSH Terms: conditions — Spondylarthritis; Radiculopathy | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Study Group will be receiving a nutraceutical product daily, for 3 months,
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Study Group will receive 10 sessions of rehabilitation program and nutraceutical product daily for 3 months.
  Interventions: Combination Product: All patients in the study will be included in rehabilitation program; Dietary Supplement: Study Group will receive a nutraceutical product daily, 3 months.
- Control Group (Active Comparator): Control Group will receive 10 sessions of rehabilitation program.
  Interventions: Combination Product: All patients in the study will be included in rehabilitation program

INTERVENTIONS:
Combination Product: All patients in the study will be included in rehabilitation program — A total of 110 consecutive participants with previous diagnosed CR lasting more than 3 months will be enrolled in this study. After initial assessment, participants without surgical recommendation, will be included into two groups: Study Group will be received 10 sessions of rehabilitation program and nutraceutical product daily, 3 months, and Control Group will be received 10 sessions of rehabilitation program. The rehabilitation program include physical therapy (electrical muscle stimulation of the neck muscle and upper limb muscles , low-Level Laser Therapy and ultrasound) and kinetic training.
Dietary Supplement: Study Group will receive a nutraceutical product daily, 3 months. — Study Group will receive a nutraceutical product daily, 3 months in addition to the rehabilitation program.
  Arms: Study Group

SUMMARY:
The investigators perform a prospective controlled study and analyse the effects of a rehabilitation program, including oral anti-inflammatory drugs, nutraceutical - ProHumano+ SpineDinamic (PHSD), physical therapy and kinetic measures on reduction of the severity of radicular pain, and improvement of the quality of life in participants with cervical radiculopathy (CR) over a relatively short period of treatment (three months).

The major tasks in the assessment and management of CR are to exclude signs and/or symptoms of possible serious underlying pathology, to focus on an active approach to promote the natural recovery and to prevent chronicity through early tailored rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* patients older than 50 years of age;
* lasting more than 3 months and diagnosed with CR confirmed by MRI in the last 6 months;
* absence of other significant and disability upper limb osteoarthritis;
* patients with stable cardiovascular and respiratory function, without unstable medical conditions;
* compliance with physical exercise during the healthcare program.

Exclusion Criteria:

* pregnancy or breastfeeding;
* need for surgical treatment;
* intolerance to any component of the nutraceutical product;
* malignancy;
* modified laboratory test (ALT, AST, or Urea >2x% reference range, Creatinine >3x% reference range).

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 3 months
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Score: /50 Transform to percentage score x 100 = %points Scoring: For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated Minimum Detectable Change (90% confidence): 5 points or 10 %points
Visual Analogue Scale For Pain | 3 months
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. Values close to 100 show a maximum value of pain, and 0 the absence of pain.

SECONDARY OUTCOMES:
Improving quality of life- Katz Index of Independence in Activities of Daily Living | 3 months
  The Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL, is the most appropriate instrument to assess functional status as a measurement of the participants ability to perform activities of daily living independently. Investigators typically use the tool to detect problems in performing activities of daily living and to plan care accordingly. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Participants are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Diana Kamal, Craiova, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR